CLINICAL TRIAL: NCT01118234
Title: International, Multicentre, Randomized Phase III Study of Rituximab as Maintenance Treatment Versus Observation Alone in Patients With Chronic Lymphocytic Leukemia
Brief Title: Rituximab Versus Observation as Maintenance Therapy in Chronic Lymphocytic Leukemia (Chronic Lymphocytic Leukemia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mabtenance
Record Dates: First submitted 2010-05-03; First posted 2010-05-06 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Rituximab; Maintenance
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental): Treatment with Rituximab 375 mg/m² every 3 months for 24 months
  Interventions: Drug: Rituximab
- Observation (No Intervention): Observation for 24 months

INTERVENTIONS:
Drug: Rituximab — Rituximab (MabThera, F. Hoffmann-La Roche Ltd., Basel, Switzerland) 375 mg/m² every 3 months for 24 months (8 infusions) or observation
  Arms: Rituximab

SUMMARY:
The purpose of the study is to evaluate the ability of Rituximab maintenance therapy to prolong progression free survival in patients with chronic lymphocytic leukemia, who responded to a Rituximab induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* B-CLL
* Age >18
* ECOG performance status 0-2
* Previous Rituximab containing induction treatment of the CLL in 1st or 2nd line
* Patient must be in complete remission or partial remission after an induction treatment containing rituximab
* ANC (absolute neutrophil count) > 1,0 x 10e9 /L
* Life expectancy > 6 months
* Patient´s written informed consent
* Patient using a reliable means of contraception for the duration of the treatment including 2 months thereafter

Exclusion Criteria:

* Active uncontrolled bacterial, viral or fungal infection
* Significantly reduced organ functions and bone marrow dysfunction not due to CLL
* creatinine clearance of below 30mL/min
* Patients with a history of other malignancies within 2 years prior to study entry
* Patients with a history of severe cardiac disease
* Other known comorbidity with the potential to dominate survival
* Transformation to aggressive B-cell malignancy
* Hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the applied drugs
* Medical condition requiring prolonged (> 1 month) use of oral corticosteroids
* Pregnant or breast feeding women
* Any coexisting medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
progression free survival | 48 months
  Clinical PFS is defined as the period from randomization until disease progression according to the NCI criteria or death due to the underlying disease.

SECONDARY OUTCOMES:
MRD (minimal residual disease) progression free survival | 48 months
  Minimal residual disease progression-free survival is defined as the period from randomization until increase of MRD levels in peripheral blood above 10-3 or, if above 10-3 before, increase of one common logarithm.
conversion rate to MRD negative | 48 months
median MRD levels | 48 months
conversation rate to CR | 48 months
effect of MRD levels on clinical PFS and OS | 48 months
event free survival | 48 months
time to next treatment | 48 months
overall survival | 48 months
Safety of Rituximab maintenance treatment in patients with CLL | 48 months
  All grades of infections and G3/4 other clinical adverse events will be documented using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0
benefit according to cytogenetic risk group (trisomy 12, del 11q, del 17p and del 13q), IgVH mutation status, ZAP 70 and CD38 expression | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof. Dr., Principal Investigator — Arbeitsgemeinschaft medikamentoese Tumortherapie
Locations (22):
- Austria (11):
  - Landesklinikum Krems, Hämato-onkologisches Service, Krems, Lower Austria
  - A.ö. Bezirkskrankenhaus Hall in Tirol, Innere Medizin / Hämato - Onkologie, Hall in Tirol, Tyrol
  - Universitätsklinik Innsbruck, Innere MEdizin IV / Hämato-Onkologie, Innsbruck, Tyrol
  - A.ö. Bezirkskrankenhaus Kufstein, Innere Medizin / Hämatologie / Onkologie, Kufstein, Tyrol
  - AKH Linz, Department für Innere Medizin 3, Linz, Upper Austria
  - Landeskrankenhaus Steyr, Innere Medizin, Hämatologie, Onkologie, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Abteilung für Innere Medizin IV, Wels, Upper Austria
  - LKH Feldkirch, Interne E, Feldkirch, Vorarlberg
  - Universitätsklinik der PMU Salzburg, Univ-Klinik für Innere Medizin, Salzburg
  - AKH Wien, Klinische Abteilung für Hämatologie und Hämostaseologie, Vienna
  - Hanusch Krankenhaus, 3. Med. Abtlg., Vienna
- Czechia (5):
  - FN Brno, Brno
  - FN Hradec Kralove, Hradec Králové
  - FN Olomouc, Olomouc
  - FN Kralovske Vinohrady, Prague
  - VFN Praha 2, Prague
- Slovakia (6):
  - F.D. Rossevelt hospital, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
  - FNsP sv. Cyrila a Metoda, Bratislava
  - FNsP L.Pasteura, Košice
  - Martinska fakultna nemocnica, Martin
  - FNsP J.A. Reimana, Prešov

REFERENCES:
- [Derived] Greil R, Obrtlikova P, Smolej L, Kozak T, Steurer M, Andel J, Burgstaller S, Mikuskova E, Gercheva L, Nosslinger T, Papajik T, Ladicka M, Girschikofsky M, Hrubisko M, Jager U, Fridrik M, Pecherstorfer M, Kralikova E, Burcoveanu C, Spasov E, Petzer A, Mihaylov G, Raynov J, Oexle H, Zabernigg A, Flochova E, Palasthy S, Stehlikova O, Doubek M, Altenhofer P, Pleyer L, Melchardt T, Klingler A, Mayer J, Egle A. Rituximab maintenance versus observation alone in patients with chronic lymphocytic leukaemia who respond to first-line or second-line rituximab-containing chemoimmunotherapy: final results of the AGMT CLL-8a Mabtenance randomised trial. Lancet Haematol. 2016 Jul;3(7):e317-29. doi: 10.1016/S2352-3026(16)30045-X. Epub 2016 Jun 16. PMID 27374465